CLINICAL TRIAL: NCT01750242
Title: OPTIVISE Map Concordance Study in DBS for Parkinson's Disease
Brief Title: Retrospective, Non-significant Risk, Deep Brain Stimulation (DBS) Care Management Software Feasibility Study
Acronym: DBS
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1669
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinson's disease Subjects: Subjects with advanced Parkinson's Disease implanted with Medtronic DBS system in the subthalamic nucleus (STN).
  Interventions: Device: Medtronic DBS system

INTERVENTIONS:
Device: Medtronic DBS system — Advanced Parkinson's disease patients implanted with the Medtronic Deep Brain Stimulation (DBS) system.

SUMMARY:
To evaluate DBS device settings and match with the features of the DBS care management software.

DETAILED DESCRIPTION:
This is a study done on Parkinson disease subjects who have received the DBS system implanted in their subthalamic nucleus.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Medtronic Deep Brain Stimulation therapy for idiopathic levodopa responsive Parkinson's Disease
* Patient who has had lead placement in the Subthalamic nucleus
* Patient with pre-op MRI available
* Patient with post-op CT scan available showing placement of the lead
* Patient who has documented improvement of at least 35% on UPDRS III scores from baseline preoperative off medication state compared to post DBS implant stimulation on/medications off

Exclusion Criteria:

* Patient who has had clinically significant persistent stimulation related adverse effects
* Patient who has evidence of lead migration without lead revision
* Patient with other brain malformations that would make it difficult to process images (ablative surgery in the basal ganglia, resective surgery, brain tumor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients who have been implanted with the DBS system
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Pahwa, MD, Principal Investigator — Parkinson's Disease and Movement Disorder Center, University of Kansas Medical Center; Melissa Houser, MD, Principal Investigator — Scripps Clinic Division of Neurology
Locations (2):
- United States (2):
  - Scripps Clinic, Division of Neurology, La Jolla, California
  - Parkinson's Disease and Movement Disorder Center, University of Kansas Medical Center, Kansas City, Kansas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following enrollment but prior to analysis, MRIs were evaluated for readability. Those unreadable were excluded from analysis (N=3).
Groups:
- PD Patients Implanted With DBS System: Subjects implanted with Medtronic DBS system for the treatment of Parkinson's disease with leads in the subthalamic nucleus who consented for the study.
Period: Overall Study
Arm/Group | PD Patients Implanted With DBS System
Started | 23
Readable Images | 20 (Subjects with readable images were analyzed and there were 3 subjects with unreadable images.)
Completed | 20
Not Completed | 3
Not completed — Unreadable Images | 3

BASELINE CHARACTERISTICS:
Population: Per protocol
Groups:
- Subjects With Advanced Parkinson's Disease: Subjects with advanced Parkinson's Disease implanted with Medtronic DBS system and with documented improvement of at least 35% on UPDRS III from baseline preoperative off medication to post-DBS implant stimulation on/medication off.
Arm/Group | Subjects With Advanced Parkinson's Disease
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
UPDRS III scores at baseline [Mean (Standard Deviation); unit: units on a scale] — Patients with documented improvement of UPDRS III scores of at least 35% were included in the study. A higher score means more motor dysfunction. The score can range from 0 -108.
  units on a scale | 39.4 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: To Characterize the Percentage of Leads in Which the Target Map and the Clinically-derived Activation Map Overlap
Description: The one-sided 95% exact binomial lower confidence bound of the proportion was calculated from subjects with readable images enrolled in the study.
Time Frame: 18 months
Population: Per Protocol
Measure: Number; unit: percentage of leads
Units Other Than Participants: leads
Groups:
- PD Patients Implanted With DBS System: Subjects implanted with Medtronic DBS system for the treatment of Parkinson's disease with leads in the subthalamic nucleus and with readable images.
Arm/Group | PD Patients Implanted With DBS System
Number analyzed (Participants) | 20
Number analyzed (leads) | 37
percentage of leads | 86.5
Statistical Analysis 1: Comparison: PD Patients Implanted With DBS System; A 95% lower confidence bound was calculated on the percentage of leads where an overlap existed. A subject may have 1 or 2 leads included in the analysis; Test type: Superiority or Other; % of leads = 86.5, 95% CI 1-sided [lower limit 73.7]

2. Secondary Outcome: Additional Study Measure on Unified Parkinson's Disease Rating Scale (UPDRS) III Scores
Description: The summary of UPDRS III medication off score at baseline and the UPDRS III stimulation on/medication off score at follow-up and the change from baseline to 18 months. The UPRS III has a range of 0 - 108.
Time Frame: Change from baseline to 18 months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects With Advanced Parkinson's Disease
Number analyzed (Participants) | 20
units on a scale | -22.5 (8.7)
Statistical Analysis 1: Comparison: Subjects With Advanced Parkinson's Disease; Summary statistics on the UPDRS III score. A higher score is more motor dysfunction; Test type: Superiority or Other; Mean Difference (Net) = -22.5, 95% CI 2-sided [-26.5 to -18.4], Standard Deviation 8.7

ADVERSE EVENTS:
Time Frame: No safety data collected
Description: The protocol for the study did not include safety data collection
Groups:
- Subjects With Advanced Parkinson's Disease: The study protocol did not require safety data to be collected for the study.
Arm/Group | Subjects With Advanced Parkinson's Disease
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less